CLINICAL TRIAL: NCT02705118
Title: Evaluation of Performance of S-fusion for Radiofrequency Ablation of Hepatocellular Carcinoma: A Randomized, Prospective Study
Brief Title: Evaluation of Performance of Automatic Fusion for Radiofrequency Ablation of Hepatocellular Carcinoma
Acronym: FAME-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JOON-IL CHOI (Other)
Responsible Party: Sponsor-Investigator, JOON-IL CHOI, Associate professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC15DNSI0039
Record Dates: First submitted 2015-12-15; First posted 2016-03-10 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: radiofrequency ablation; image fusion
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automatic registration arm (Experimental): Automatic registration for fusion imaging of US and MRI will be performed.
  Automatic Imaging fusion of ultrasonography and MRI
  Interventions: Device: Automatic Imaging fusion of ultrasonography and MRI
- Manual registration arm (Active Comparator): Manual registration for fusion imaging of US and MRI will be performed.
  Manual Imaging fusion of ultrasonography and MRI
  Interventions: Device: Manual Imaging fusion of ultrasonography and MRI

INTERVENTIONS:
Device: Automatic Imaging fusion of ultrasonography and MRI — Radiofrequency ablation for hepatic malignancies will be performed with automatic registration registration. Except the imaging registration, all other procedures for RF ablation is same.
  Arms: Automatic registration arm
Device: Manual Imaging fusion of ultrasonography and MRI — Radiofrequency ablation for hepatic malignancies will be performed with manual registration registration. Except the imaging registration, all other procedures for RF ablation is same.
  Arms: Manual registration arm

SUMMARY:
Fusion imaging of US and MRI is very helpful for interventional procedure such as radiofrequency ablation in liver. However, manual registration of US and magnetic resonance (MR) imaging is somewhat time-consuming and difficult for less-experienced physicians. Recently, automatic registration function was developed to help the fusion of US and CT/MRI imaging. The purpose of this trial is to compare the registration time and accuracy of manual registration system and automatic registration system.

DETAILED DESCRIPTION:
1. Patients will be randomized and assigned.
2. For automatic registration group, automatic image fusion will be done by RS80A US unit and RF ablation will be performed. Image fusion time will be measured.
3. For manual registration group, manual image fusion will be done by LOGIQ-E9 US unit and RF ablation will be performed. Image fusion time will be measured.

3) After radiofrequency (RF) ablation, immediate, contrast enhanced CT will be performed to evaluate technical success and complications 4) Accuracy of registration will be measured by home-made software using 3D techniques.

5) After one month, technical effectiveness will be evaluated by contrast enhanced CT 6) F/U of CT images will be obtained until one year after RF ablation with a interval of 1-3 months.

ELIGIBILITY:
Inclusion Criteria:

* More than 40-years old
* Patients with hepatic malignancy who will underwent radiofrequency ablation

Exclusion Criteria:

* Not using fusion imaging (CT guidance or fluoroscopic guidance)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Registration accuracy | Immediately after RF ablation
  Accuracy of imaging fusion (US and MRI)

SECONDARY OUTCOMES:
Technical success | Within 48 hours after RF ablation
  Completeness of tumor ablation
Technical effectiveness | One month after RF ablation
  Completeness of tumor ablation
Registration time | Within 48 hours after RF ablation
  Time required for registration

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Il Choi, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No